CLINICAL TRIAL: NCT06012357
Title: Nociception Coma Scale-Revised Recorded After Personalized Stimulus May Improve Assessment of Pain Responses in Non-communicative Patients With Disorders of Consciousness. An International Multicentric Study
Brief Title: Pain Protocol: Nociception Coma Scale-Revised With Personalized Stimulus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Rita Formisano, Director of Neuroriabilitazione 2, I.R.C.C.S. Fondazione Santa Lucia
Other Study IDs: CE/PROG.603
Record Dates: First submitted 2023-04-07; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Disorder of Consciousness
Keywords: Disorder of consciousness; Pain; Responsiveness; Nociception Coma Scale-Revised; Coma Recovery Scale-Revised; Non communicative patients
MeSH Terms: conditions — Consciousness Disorders; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nociception Coma Scale-Revised — Nociception Coma Scale-Revised Recorded after personalized painful stimulus

SUMMARY:
The goal of this observational study is to compare Nociception Coma Scale-Revised Recorded (NCS-R) scores obtained with the standard pressure on fingernail bed (standard stimulus, SS) versus other personalized painful stimuli (PS), in non-communicative patients with disorders of consciousness (DoC), as indicated by professionals and caregivers involved in their care and rehabilitation. The study aims also to establish possible correlations between NCS-R and Coma Recovery Scale-Revised (CRS-R.) The main question : an integrated patient-centered approach for assessment of the physical pain, in which clinical measures and behavioral observations will be integrated, to understand and manage the pain intensity, may improve treatment and rehabilitation outcome. Specifically, a new version of NCS-R, adapted with PS, may produce more intentional and specific responses to pain-inducing maneuvers. Investigating pain perception in non-communicative patients, through recognition of a personalized source of nociception and pain, may avoid non specific, useless and harmful noxious tests (as with standard pain scales) and may provide tools for revealing nociception even in the lack of any response to standard clinical evaluation.

Question 1: the superiority of personalized painful stimulus a standard painful stimulation in nin communicative patients.

Question 2: the parallel recovery of painful stimuli responsiveness and consciousness Participants will Responsiveness and pain perception will be assessed respectively with the CRS-R and the NCS-R. Pain responses will be assessed by means of standard stimulus (NCS-R-SS, as used in the CRS-R) and personalized stimulation (NCS-R-PS), at admission and discharge.

CRS-R will be administered within the first month after admission, at least 5 times in different days, choosing the highest score as reference and repeated during recovery of consciousness or discharge.

After informed consent by patient's legal representative or the primary caregiver, for the purpose of the study, caregivers (including relatives, nurses, therapists, physicians) will be asked to record all manoeuvres they feel are associated with potential pain, with a window of observation of the rehabilitation and nursing staff of around one week to identify the personalized painful stimulus (about the second week after admission at the rehabilitation ward). Amongst them, the manoeuvres that consistently over time induced the most motor/behaviour responses suggestive of pain perception, reported at least by 2 members of the rehabilitation staff or by one of them and one caregiver, will be chosen as the personalized stimulus (PS). NCS-R with standard stimulus (NCS-R-SS) and with personalized stimulus (NCS-R-PS), will be recorded within 30 days after admission, alternating the order of the 2 painful stimulations; CRS-R will be recorded accordingly, in parallel to NCS-R-SS and NCS-R-PS and will be blindly recorded, at the same time, by two different rehabilitation staff members, to assess inter-rater reliability, whereas two of them will repeat both NCS-R_SS and NCS-R-PS during the same week to assess intra-rater reliability of both NCS-R-SS and NCS-R-PS, with an interval of at least 6 hours from the last pain killer or anti-spastic drugs administration, including GABAergic, anti-inflammatory drugs or opiates.

Both CRS-R and NCS-R (SS and PS) will be repeated 1 month and 3 months after the first assessment with the same procedures of the first time.

ELIGIBILITY:
Inclusion Criteria:

* severe acquired brain injury (sABI),
* clinical history and neuroimaging (brain CT and/or MRI) and fulfilling the criteria proposed for the sABI diagnosis:
* Glasgow Coma Scale (GCS) score ≤ 8 within 24 hours after injury,
* diagnosis of disorders of consciousness (DoC), (VS/UWS or MCS), according to the Coma Recovery Scale-Revised (CRS-R),
* interval from the acute event of at least 3 months.

Exclusion Criteria:

* history of previous brain injury,
* neurological or psychiatric disorders,
* alcohol or illicit drug abuse and concomitant spinal cord injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (age ≥ 18 years) diagnosed with Vegetative State (VS)/Unresponsive Wakefulness Syndrome (UWS) or Minimally Conscious State (MCS) after severe acquired brain injury (ABI) admitted to neurorehabilitation ceters.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain perception in non communicative patients | Within 30 days after admission
  Time 0

SECONDARY OUTCOMES:
Superiority of personalized painful stimulus versus standard stimulation | 30 days from T0
  Time 1

OTHER OUTCOMES:
Possible parallel recovery of painful stimulus responsiveness and consciousness | 3 months from T0
  Time 2

CONTACTS AND LOCATIONS:
Locations (1):
- Rita Formisano, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Enrollment of at least 50 patients with DoC in the participating centers

REFERENCES:
- [Derived] Formisano R, Aloisi M, Ferri G, Schiattone S, Estraneo A, Magliacano A, Noe E, Perez MDN, Hakiki B, Romoli AM, Bertoletti E, Leonardi G, Thibaut A, Martial C, Gosseries O, Brisbois M, Lejeune N, O'Valle M, Ferri J, Frederick A, Zasler N, Schnakers C, Iosa M. Nociception Coma Scale-Revised with Personalized Painful Stimulus Versus Standard Stimulation in Persons with Disorders of Consciousness: An International Multicenter Study. J Clin Med. 2024 Sep 18;13(18):5528. doi: 10.3390/jcm13185528. PMID 39337015